CLINICAL TRIAL: NCT02433808
Title: Neostigmine Reversal And Neuromuscular Recovery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Endeavor Health (Other)
Responsible Party: Principal Investigator, Glenn S. Murphy, MD, Director Clinical Research, Endeavor Health
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: EH15-089
Record Dates: First submitted 2015-04-24; First posted 2015-05-05 (Estimated); Last update posted 2017-04-12 (Actual); Status verified 2017-04

CONDITIONS: Residual Neuromuscular Block
MeSH Terms: conditions — Delayed Emergence from Anesthesia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Neostigmine Group (Experimental): Neostigmine will be administered at the conclusion of the surgical procedure
  Interventions: Drug: Neostigmine Group
- No Neostigmine group (Placebo Comparator): Saline will be administered at the conclusion of the surgical procedure
  Interventions: Other: No Neostigmine group

INTERVENTIONS:
Drug: Neostigmine Group — Neostigmine will be used to reverse neuromuscular block at the conclusion of the surgical procedure. The effect on muscle strength will be determined using the TOF-Watch-SX and clinical examination
  Arms: Neostigmine Group
Other: No Neostigmine group — Saline will be administered to patients at the end of the surgical procedure when neuromuscular function has recovered
  Other Names: Placebo Comparator
  Arms: No Neostigmine group

SUMMARY:
Patients undergoing surgery often receive paralytic agents (or neuromuscular blocking agents (NMBAs)) to facilitate the procedure. At the end of surgery, the effects NMBAs are reversed with a drug called neostigmine. The use of neostigmine significantly reduces the risk that a patient will be left with muscle weakness in the recovery room. Many anesthesiologists routinely use neostigmine because postoperative muscle weakness may lead to adverse events after surgery. Other anesthesiologists do not routinely administer neostigmine in the operating room because of concerns about potential side effects. Surprisingly, some investigators have reported that neostigmine-induced muscle weakness may occur if the drug is given when the effects of the NMBAs have completely worn off. In contrast, other investigators have not observed this side effect when neostigmine was given at the end of surgery. The aim of this study is to determine whether neostigmine use is associated with muscle weakness when it is given at the time of nearly complete recovery from NMBAs. Muscle strength will be measured using a sensitive monitor (TOF-Watch-SX) and through an examination of the patient for evidence of muscle weakness. Patients will also be evaluated how they recover from anesthesia and surgery.

DETAILED DESCRIPTION:
120 patients will be enrolled in this randomized clinical trial. Patients will be assigned, via a computer-generated randomized table, to either a neostigmine group or a no neostigmine group. Patients in the neostigmine group will receive neostigmine 40 µg/kg at the end of the surgical procedure when TOF ratios have recovered to 0.9 or greater. Patients in the no neostigmine group will be administered saline (control) at the time of neuromuscular recovery. Patients with TOF ratios < 0.9 will be excluded from either study cohort. These subjects will be administered neostigmine 50 µg/kg at the conclusion of surgery. The same postoperative data (see below) will be recorded in this group as will be collected in the two study cohorts in order to determine the characteristics of patients not achieving spontaneous recovery.

Anesthetic care will be standardized in both study groups. Patients will be induced with propofol 1-2 mg/kg, fentanyl 100 µg/kg, and rocuronium as the NMBA (1 X ed 95 dose). No further rocuronium will be administered unless requested by the surgeon. Clinicians will be instructed to manage neuromuscular blockade so that full recovery of muscle strength is present at the end of the surgical procedure.

Neuromuscular blockade in the operating room will be quantified with the TOF-Watch-SX, an FDA-approved quantitative monitoring device. After induction of anesthesia, baseline data will be collected. A 5-second 50 Hz tetanic stimulation will be applied to reduce the time required to achieve baseline signal stabilization. After signal stability is achieved, the TOF-Watch will be calibrated and then a baseline TOF value recorded. Rocuronium will then be administered and the oral endotracheal tube placed 2-4 minutes later. Neuromuscular blockade will be managed to allow spontaneous recovery of neuromuscular function to occur, with the goal of reaching a TOF ratio of ≥ 0.9 at the end of the surgical procedure. At the time when neostigmine is typically administered, one of two syringes will be attached to the intravenous line, and the clear solution (neostigmine or saline) given. These syringes will be prepared prior to the end of surgery. For patients in the in the neostigmine group, 40 µg/kg of neostigmine (with an appropriate dose of glycopyrrolate) will be drawn up into the syringe and labeled accordingly. For patients in the no neostigmine group, an equal volume of saline will be drawn into a syringe, and a neostigmine label applied to the syringe. Both the neostigmine and saline solutions are clear and indistinguishable (to be prepared by pharmacy). Thereafter, all data collection will be obtained by research assistants blinded to group assignment.

Immediately prior to neostigmine or saline administration, TOF ratios will be recorded, and then the syringe attached to the intravenous line and the solution injected. Train-of-four ratios will then be recorded every 12 seconds until the time of tracheal extubation.

During transport from the operating room to the PACU, a research assistant will observe oxygen saturation levels, and the lowest value recorded. Oxygenation by pulse oximeter will also be monitored and recorded for the first 30 minutes of the PACU admission (every 1 minute via the PACU monitoring system). The need for addition oxygen therapy at any time following extubation will be noted. During this same time period (from extubation until 30 minutes after the PACU arrival) patients will be carefully observed for any evidence of airway obstruction or need for maneuvers to maintain a patent airway. This data will be recorded by the research assistant and the PACU nursing staff. In addition, 15 minutes after the PACU admission, subjects will be examined for 11 signs and 16 symptoms of muscle weakness. This examination will be performed by the blinded research assistant. The times required to achieve discharge criteria and actual PACU discharge will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Ages of 18-80
* Patients undergoing general anesthesia requiring endotracheal intubation
* Procedures that do not require maintenance of neuromuscular blockade for completion of the surgical procedure

Exclusion Criteria:

* Presence of renal failure (creatinine > 2.0 mg/dL)
* Neuromuscular disease impacting upper airway musculature or neuromuscular monitoring
* Lack of access to either upper extremity for monitoring
* Procedure duration less than 30 minutes
* Requirement for postoperative intubation
* Patients not achieving a TOF ratio of ≥ 0.9 at the end of surgery will be excluded from either study cohort.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Change in train-of-four (TOF) ratio | 30 minutes after the end of the surgical procedure
  The effect of neostigmine or placebo (saline) on TOF ratios, when given at full neuromuscular recovery, will be assessed

SECONDARY OUTCOMES:
airway obstruction-presence or absence (yes or no) | 30 minutes after the end of the surgical procedure
  Any episodes of airway obstruction will be recorded
hypoxemic events (oxygen saturation by pulse oximeter (SpO2) < 94%) | 30 minutes after the end of the surgical procedure
  Any hypoxemic events will be recorded

CONTACTS AND LOCATIONS:
Locations (1):
- NorthShore University HealthSystem, Evanston, Illinois, United States